CLINICAL TRIAL: NCT04106856
Title: SHAPER: A Phase 1 Study of Losartan and Hypofractionated Radiation Therapy After Induction Chemotherapy for Borderline Resectable or Locally Advanced Pancreatic Cancer
Brief Title: Losartan and Hypofractionated Rx After Chemo for Tx of Borderline Resectable or Locally Advanced Unresectable Pancreatic Cancer (SHAPER)
Acronym: SHAPER
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI121104; NCI-2019-05882 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCI121104 (Other: Huntsman Cancer Institute/University of Utah); P30CA042014 (NIH)
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Borderline Resectable Pancreatic Adenocarcinoma; Locally Advanced Pancreatic Ductal Adenocarcinoma; Locally Advanced Unresectable Pancreatic Adenocarcinoma; Stage II Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8; Stage IIB Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiation Dose Hypofractionation; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (losartan, hypofractionated radiation therapy) (Experimental): Beginning on day 1, patients receive losartan potassium PO QD. Beginning day 14, patients also undergo hypofractionated radiation therapy over 15 fractions 5 days a week for up to 3 weeks. Patients continue to receive losartan potassium PO QD during radiation therapy and for 28 days after completion of radiation therapy. Patients may begin additional anti-cancer therapy per investigator discretion after the last dose of HRT. Losartan can be given concurrently with additional therapy and Losartan dosing can continue until 28 days after last dose of HRT, regardless of when additional therapy is started.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Drug: Losartan; Drug: Losartan Potassium; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation
Drug: Losartan — Given PO
Drug: Losartan Potassium — Given PO
  Other Names: Cozaar; losartan
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects of losartan and hypofractionated radiation therapy after chemotherapy in treating patients with pancreatic cancer that may or may not be removed by surgery (borderline resectable) or has spread from its original site of growth to nearby tissues or lymph nodes and is not amenable to surgical resection (locally advanced unresectable). Losartan may improve blood flow and allows for better tissue oxygenation. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Giving losartan and hypofractionated radiation therapy may work better in treating patients with pancreatic cancer compared to hypofractionated radiation therapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety of losartan potassium (losartan) in combination with hypofractionated radiation treatment for patients with stable or locally progressive pancreatic ductal adenocarcinoma (PDAC) after induction chemotherapy.

SECONDARY OBJECTIVES:

I. To assess the safety of losartan in combination with HRT for patients with stable or locally progressive PDAC after induction chemotherapy.

II. To assess the efficacy of losartan in combination with HRT for patients with stable or locally progressive PDAC after induction chemotherapy.

III. To assess the rate of hypotensive adverse events grade >= 3.

EXPLORATORY OBJECTIVE:

I. To assess patient reported quality of life.

OUTLINE:

Beginning day 1, patients receive losartan potassium orally (PO) once daily (QD). Beginning day 14, patients also undergo hypofractionated radiation therapy over 15 fractions 5 days a week for up to 3 weeks. Patients continue to receive losartan potassium PO QD during radiation therapy and for 28 days after completion of radiation therapy.

After completion of study treatment, patients are followed up at 28 and 84 days, every 3 months for 12 months, and then every 6 months for up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pancreatic ductal adenocarcinoma
* Borderline resectable or locally advanced unresectable pancreas cancer as defined by the National Comprehensive Cancer Network (NCCN) and determined by a pancreatic surgeon prior to therapy. This can be confirmed by the surgeon?s documentation in the electronic medical record, by a treatment planning conference note, or by the signature of a pancreatic surgeon
* At least one infusion of FOLFIRINOX, NALIRIFOX, or gemcitabine based chemotherapy must have been attempted.
* No more than 6 months of chemotherapy as defined by standard cycle lengths (every other week infusions for FOLFIRINOX or NALIRIFOX, and 3 infusions per month for gemcitabine-based therapy). Each infusion of FOLFIRINOX or NALIRIFOX will be counted as 0.5 months. Three infusions of gemcitabine based chemotherapy will be counted as 1 month. If chemotherapy is given over a protracted period, then more than 6 months of chemotherapy may be acceptable. For example, if gemcitabine-based therapy is given every other week, then each infusion will still only count as 1/3 of a month toward the 6 month total. If a partial cycle of chemotherapy is given, that partial cycle will be counted proportional to the amount given. For example, if one of three planned infusions of gemcitabine based chemotherapy is given, it will be counted as 1/3 month.
* Enrollment must occur within 90 days of Day 1 of the last infusion given of chemotherapy. Patients who have primary tumor or regional lymph node progression on chemotherapy or prior to enrollment are eligible if no distant metastases are identified on the screening imaging assessment.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelets >= 100k/uL
* Total Bilirubin =< 2.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN)
* Serum creatinine < 1.25 md/dL
* Serum potassium < 5.0 mmol/L
* Negative serum or urine pregnancy test at screening for women of childbearing potential
* Highly effective contraception for both male and female subjects throughout the study and for at least 12 months after last study treatment administration if the risk of conception exists
* Recovery to baseline or =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) v5.0 from toxicities related to any prior treatments, unless AEs are clinically nonsignificant and/or stable on supportive therapy
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines

Exclusion Criteria:

* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen of this trial
* Distant metastases. Regional lymphatic disease is acceptable
* Prior radiation therapy or definitive resection for pancreatic cancer
* Uncontrolled gastric or duodenal ulcer disease within 28 days of registration
* Chronic cough, defined 30% of days over 3 months with active symptoms at enrollment or over 12 months with last active symptoms occurring 6 months prior to enrollment
* Symptomatic hypotension (blood pressure < 90 systolic or < 60 diastolic at screening vital sign assessment) that has the potential to interfere with the patient's safety or ability to complete protocol treatment, at the discretion of the treating investigator
* Patients taking > 50mg losartan QD who, at the discretion of the treating investigator, cannot be reduced to the protocol defined regimen.
* Patients taking an angiotensin II receptor blocker or an angiotensin-converting enzyme inhibitor who, at the discretion of the treating investigator, cannot be safely discontinued prior to Day 1 dosing.
* Patients taking direct renin-angiotensin system inhibitors including aliskiren (Rasilez).
* Prior allergy to an angiotensin II receptor blocker
* Concurrent use of direct renin inhibitor including aliskiren (Rasilez)
* Patients with known history of:

  * Heart failure. Patients with heart failure, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
  * Patients with a prior history of treatment with cardiotoxic agents should be evaluated for heart failure prior to enrollment at the discretion of the treating investigator.
  * Solitary kidney, renal artery stenosis, or chronic renal failure
* Human immunodeficiency virus (HIV)-infected patients who are not on effective anti-retroviral therapy or have a detectable viral load within 6 months of trial entry
* Patients with known evidence of chronic hepatitis B virus (HBV) infection and a detectable HBV viral load
* Patients with a history of hepatitis C virus (HCV) infection who have not been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Subject is currently enrolled on another investigational treatment study for pancreas cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2026-08-08 (Estimated)

PRIMARY OUTCOMES:
Grade 3 or higher gastrointestinal toxicity rate | Up to 3 months (84 days) after completion of radiation therapy
  Will be graded according to Common Terminology Criteria for Adverse Events version (v) 5.0. The proportion of subjects that experience this endpoint will be tabulated along with an exact 90% binomial confidence interval (Clopper-Pearson).

SECONDARY OUTCOMES:
Frequency of adverse events | Up to 3 months (84 days) after completion of radiation therapy
  Will be graded according to Common Terminology Criteria for Adverse Events version (v) 5.0.
Response rate (clinical and/or pathologic partial response [PR] and complete response [CR]) | Up to 36 months post-treatment
  Will be described using Response Evaluation Criteria in Solid Tumors v1.1. The proportion of subjects with a PR and CR will be reported along with exact binomial confidence intervals (Clopper-Pearson).
Progressive free survival (PFS) | From the time of enrollment until disease progression or death (any cause), assessed up to 36 months post-treatment
  Kaplan-Meier methods will be used to report PFS.
Overall survival (OS) | From the patient?s first dose of study drug to death due to any cause, assessed up to 36 months post-treatment
  Kaplan-Meier methods will be used to report OS.
Number patients that require a medical intervention or hospitalization due to hypotension | Up to 36 months post-treatment
  Will be analyzed descriptively.

OTHER OUTCOMES:
Patient reported quality of life assessment- review of symptoms and how they interfere in life | At study entry, during the final week of radiation therapy, and at each follow up visit
  Will be assessed using MD Anderson Symptom Inventory-Gastrointestinal (MDASI-GI).

CONTACTS AND LOCATIONS:
Overall Officials: Shane Lloyd, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No